CLINICAL TRIAL: NCT03489538
Title: Homocysteine After Laparoscopic Roux-enY Gastric Bypass: a Comprehensive Evalutation in 708 Patients
Brief Title: Homocysteine After Laparoscopic Roux-enY Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Prager, associate professor, MD, Medical University of Vienna
Other Study IDs: EK1143
Record Dates: First submitted 2018-02-22; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Morbid; Homocystine; Metabolic Disorder; Bariatric Surgery Candidate; Folate Deficiency; Vitamin B 12 Deficiency
Keywords: bariatric surgery; gastric bypass; homocysteine; folate; vitamin b12
MeSH Terms: conditions — Obesity, Morbid; Metabolic Diseases; Folic Acid Deficiency; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Collection of blood samples during routine pre- and postoperative visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RYGB Patients: Laparoscopic long limb roux-en-Y gastric bypass group. All consecutive patients eligible for bariatric surgery.
  Interventions: Procedure: laparoscopic long limb roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: laparoscopic long limb roux-en-Y gastric bypass — standard laparoscopic roux-en-Y gastric bypass (biliopancreatic limb 40 to 60 cm, alimentary limb 150 cm)

SUMMARY:
Changes in homocysteine values after bariatric surgery remain controversially discussed. This is the first comprehensive summary to depict timeline changes in homocysteine levels following laparoscopic roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
Homocysteine is an independent risk factor for cardiovascular disease. Changes in homocysteine levels following bariatric surgery remain controversially discussed.

708 consecutive patients underwent laparoscopic roux-en-Y gastric bypass over a 6 year period. Throughout their routine follow-up, demographic data as well as homocysteine, folate and vitamin B12 were retrospectively collected at the timepoints: preoperatively, at 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, and 96 months postoperatively.

In order to reveal clinical relevance of the results, patients were sent a special questionnaire accompanied by an informed consent form for participation and asked for cardiovascular disease events (myocardial infarction, stroke, deep venous thrombosis) or any other hospital stay after the surgery and cross checked with two region wide databases which account for approx. 80% of all hospital contacts in the region. Additionally, the database was networked with the statewide death registry in order to reveal deceased subjects and data about their demise through the beforementioned databases was collected.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40kg/m2 or BMI > 35 kg/m2 including relevant comorbidities
* Age between 18 to 75 years
* suitable for operation, consent
* no contraindications for the operation

Exclusion Criteria:

* BMI < 35 kg/m2
* age below 18 or above 75 years
* not able to consent to the operation
* severe medical conditions not applicable for general anaesthesia
* non compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients eligible for bariatric surgery according to the american society of metabolic and bariatric surgery criteria.
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Homocysteine in µmol/l assessed by CMIA technique. | timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively
  Measured by Chemiluminescent microparticle immunoassay (CMIA) technique in µmol/l.
  Change of homocysteine over the timeframe at the timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively.

SECONDARY OUTCOMES:
Weight in kg measured by a standard scale. | timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively
  Change of weight in kg over the timeframe at the timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively.
Folate in nmol/l assessed by ELCIA method. | timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively
  ELCIA: electrochemiluminescent immunoassay Change of folate in nmol/l over the timeframe at the timepoints preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively.
Vitamin B12 in pmol/l assessed by CMIA technique. | timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively
  Change of vitamin B12 in pmol/l over the timeframe at the timepoints preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively.
Number of cardiovascular events assessed by a questionnaire and cross checking with 2 state wide databases. | Through study attendance the specific date of the incident was assessed and assigned to the timepoints: preoperatively, 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, and 96 months postoperatively
  Assessed conditions: events of myocardial infarction, stroke, deep vein thrombosis and peripheral artery disease which were not preexistent.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, MD, Principal Investigator — Medical University of Vienna, Department of Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers yet.

REFERENCES:
- [Result] Clarke R, Daly L, Robinson K, Naughten E, Cahalane S, Fowler B, Graham I. Hyperhomocysteinemia: an independent risk factor for vascular disease. N Engl J Med. 1991 Apr 25;324(17):1149-55. doi: 10.1056/NEJM199104253241701. PMID 2011158
- [Result] Williams DB, Hagedorn JC, Lawson EH, Galanko JA, Safadi BY, Curet MJ, Morton JM. Gastric bypass reduces biochemical cardiac risk factors. Surg Obes Relat Dis. 2007 Jan-Feb;3(1):8-13. doi: 10.1016/j.soard.2006.10.003. Epub 2006 Dec 27. PMID 17196442
- [Result] Woodard GA, Peraza J, Bravo S, Toplosky L, Hernandez-Boussard T, Morton JM. One year improvements in cardiovascular risk factors: a comparative trial of laparoscopic Roux-en-Y gastric bypass vs. adjustable gastric banding. Obes Surg. 2010 May;20(5):578-82. doi: 10.1007/s11695-010-0088-0. Epub 2010 Feb 26. PMID 20186576
- [Result] Borson-Chazot F, Harthe C, Teboul F, Labrousse F, Gaume C, Guadagnino L, Claustrat B, Berthezene F, Moulin P. Occurrence of hyperhomocysteinemia 1 year after gastroplasty for severe obesity. J Clin Endocrinol Metab. 1999 Feb;84(2):541-5. doi: 10.1210/jcem.84.2.5476. PMID 10022413
- [Result] Dixon JB, Dixon ME, O'Brien PE. Elevated homocysteine levels with weight loss after Lap-Band surgery: higher folate and vitamin B12 levels required to maintain homocysteine level. Int J Obes Relat Metab Disord. 2001 Feb;25(2):219-27. doi: 10.1038/sj.ijo.0801474. PMID 11410823
- [Result] Lapointe M, Poirier P, Martin J, Bastien M, Auclair A, Cianflone K. Omentin changes following bariatric surgery and predictive links with biomarkers for risk of cardiovascular disease. Cardiovasc Diabetol. 2014 Aug 21;13:124. doi: 10.1186/s12933-014-0124-9. PMID 25139582
- [Result] Sheu WH, Wu HS, Wang CW, Wan CJ, Lee WJ. Elevated plasma homocysteine concentrations six months after gastroplasty in morbidly obese subjects. Intern Med. 2001 Jul;40(7):584-8. doi: 10.2169/internalmedicine.40.584. PMID 11506296
- [Result] Toh SY, Zarshenas N, Jorgensen J. Prevalence of nutrient deficiencies in bariatric patients. Nutrition. 2009 Nov-Dec;25(11-12):1150-6. doi: 10.1016/j.nut.2009.03.012. Epub 2009 May 31. PMID 19487104
- [Result] Gomez-Ambrosi J, Pastor C, Salvador J, Silva C, Rotellar F, Gil MJ, Catalan V, Rodriguez A, Cienfuegos JA, Fruhbeck G. Influence of waist circumference on the metabolic risk associated with impaired fasting glucose: effect of weight loss after gastric bypass. Obes Surg. 2007 May;17(5):585-91. doi: 10.1007/s11695-007-9101-7. PMID 17658015
- [Result] Ledoux S, Coupaye M, Bogard C, Clerici C, Msika S. Determinants of hyperhomocysteinemia after gastric bypass surgery in obese subjects. Obes Surg. 2011 Jan;21(1):78-86. doi: 10.1007/s11695-010-0269-x. PMID 20814760
- [Result] Sledzinski T, Goyke E, Smolenski RT, Sledzinski Z, Swierczynski J. Decrease in serum protein carbonyl groups concentration and maintained hyperhomocysteinemia in patients undergoing bariatric surgery. Obes Surg. 2009 Mar;19(3):321-6. doi: 10.1007/s11695-008-9691-8. Epub 2008 Oct 2. PMID 18830787
- [Result] Tedesco AK, Biazotto R, Gebara TS, Cambi MP, Baretta GA. PRE- AND POSTOPERATIVE IN BARIATRIC SURGERY: SOME BIOCHEMICAL CHANGES. Arq Bras Cir Dig. 2016;29Suppl 1(Suppl 1):67-71. doi: 10.1590/0102-6720201600S10017. PMID 27683780

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03489538/Prot_SAP_000.pdf